CLINICAL TRIAL: NCT07098221
Title: Effects of Hydrogen-Rich Water on Resting Metabolism in Healthy Young Adults: A Randomized, Double-Blind, Placebo-Controlled Crossover Trial
Brief Title: Hydrogen-Rich Water and Resting Metabolism in Young Adults
Acronym: H2REST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Nikola Todorovic, Teaching assistant, PhD, University of Novi Sad
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 50-10-18/2024-3
Record Dates: First submitted 2025-07-17; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Healthy Subjects or Volunteers
Keywords: Hydrogen-rich water; Resting metabolism; Energy expenditure; Substrate utilization; Metabolic rate
MeSH Terms: interventions — Hydrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM1: 250 ml of Hydrogen Rich Water (Experimental): Hydrogen-producing tablets: Tablets designed to dissolve in water and release molecular hydrogen gas, creating hydrogen-rich water that can be consumed to potentially provide antioxidant and anti-inflammatory benefits.
  Interventions: Dietary Supplement: Molecular Hydrogen
- ARM 2: 250 ml of Placebo Water (Non-hydrogen-producing tablets) (Placebo Comparator): Non-hydrogen-producing tablets, identical in appearance and taste to the active supplement
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Molecular Hydrogen — Participants in this arm will consume a single 250 mL dose of hydrogen-rich water containing approximately 1.6-2.0 ppm of dissolved molecular hydrogen (H₂), The HRW will be ingested following an overnight fast, and resting metabolism will be measured approximately 30-60 minutes post-consumption using indirect calorimetry.
  Arms: ARM1: 250 ml of Hydrogen Rich Water
Dietary Supplement: Placebo Comparator — Non-hydrogen-producing tablets, identical in appearance and taste to the active supplement
  Arms: ARM 2: 250 ml of Placebo Water (Non-hydrogen-producing tablets)

SUMMARY:
The H2REST trial is a randomized, double-blind, placebo-controlled crossover study investigating the acute effects of a single dose of hydrogen-rich water (HRW) on resting metabolism in healthy young adults. Participants complete two testing sessions-receiving either HRW or placebo in a randomized order-followed by standardized metabolic testing. Primary outcomes include resting energy expenditure, respiratory exchange ratio, and substrate utilization measured via indirect calorimetry. The study aims to assess whether acute HRW intake can modulate metabolic rate and fuel preference at rest, and to explore inter-individual variability in response.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years
* BMI between 18.5 and 25.0 kg/m²
* Apparently healthy, with no history of chronic disease
* Non-smoker, not currently using nicotine-containing products
* Able to provide informed consent
* Willing to refrain from alcohol, caffeine, and strenuous exercise for 24 hours before each study visit
* Able to comply with study procedures, including fasting and attending all study visits

Exclusion Criteria:

* Diagnosed metabolic, cardiovascular, respiratory, gastrointestinal, or endocrine disorders
* Use of dietary supplements or medications affecting metabolism (within the past 2 weeks)
* Allergy or intolerance to components of the hydrogen or placebo beverages
* Pregnant or lactating
* Shift work or irregular sleep schedule
* Participation in another clinical study within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Resting Energy Expenditure (REE) | Participants will attend three study visits, with each intervention separated by a 7-day washout period to minimize carry-over effects. During each visit, measurements will be conducted approximately 30-60 minutes post-intervention.
  The measurements will be obtained during each study visit. Since this is an interventional study assessing the acute effects of molecular hydrogen, measurements will be collected three times:
  At baseline, without any intervention (pre-familiarization),
  After a single dose of molecular hydrogen, and
  After placebo administration.
  The period between each intervention will be seven days, serving as a washout period to prevent carry-over effects. All participants will be instructed to maintain their regular diet and to avoid alcohol, caffeine-containing beverages, and strenuous physical activity for at least 24 hours prior to each visit.
  Measure Type: Continuous (kcal/day)
  Method: Indirect calorimetry
  Description: To assess the effect of acute ingestion of hydrogen-rich water versus placebo on resting energy expenditure in healthy young adults.

IPD SHARING:
Plan to Share IPD: Yes